CLINICAL TRIAL: NCT02460497
Title: Multicenter, Open Label Clinical Trial to Evaluate the Effect and Tolerability of Minoxidil 2% Solution and Botanical Hair Solution Regimen in Women With Thinning Hair and Female Pattern Hair Loss/Androgenic Alopecia (Ludwig I and II)
Brief Title: Minoxidil 2% Solution and Botanical Hair Regimen in Women With Thinning Hair and Female Pattern Hair Loss/Androgenic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10330
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Female Pattern Hair Loss, Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Treatment: Minoxidil 2% / Botanical Hair Solution for Women

INTERVENTIONS:
Drug: Treatment: Minoxidil 2% / Botanical Hair Solution for Women

SUMMARY:
The purpose of this study is to characterize the effect of Minoxidil 2% Solution and Botanical Hair Solution Regimen in women with thinning hair and female pattern hair loss/androgenic alopecia (Ludwig I and II).

ELIGIBILITY:
Key Inclusion Criteria:

1. Female patients age 18 to 60 years at the time of enrollment.
2. Women who have self-perceived thinning hair.
3. Women who have presentation of female pattern hair loss/androgenic alopecia (Ludwig I and II).

Key Exclusion Criteria:

1. History of allergic reactions or severe intolerance to minoxidil and Botanical Hair Solution product ingredients.
2. Plan to use any other concomitant therapy to treat hair loss, regrowth or volume during the study.

3 Subjects taking or planning to take topical or systemic prescription or OTC medications for treating hair loss and/or hair volume.

4. Any significant history of concurrent medical disease, which in the judgment of the Investigator, would make the subject inappropriate for entry to this study including history of skin disease that may confound study results.

5. Subjects who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study.

6. Pregnant or breast-feeding females or women planning to become pregnant during the course of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2015-09-19 (Actual); Study Completion 2015-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephens & Associates, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 center in the United States from 27 May 2015 to 19 September 2015.
Pre-assignment Details: A total of 61 participants were enrolled and received treatment in this study.
Groups:
- Minoxidil 5% Foam and Botanical Hair Solution: Participant received minoxidil 2% solution 1 milliliter (1 mL) on the scalp in the hair loss area and botanical hair solution (5-10 sprays) for women on entire scalp twice per day for up to 12 weeks.
Period: Overall Study
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Started | 61
Intent-to-treat (ITT) Population | 54
Safety Population (SP) | 60
Completed | 52
Not Completed | 9
Not completed — Participant Requested Withdrawal | 4
Not completed — Non-Compliance | 1
Not completed — Did not Meet Protocol Criteria | 1
Not completed — Lost to Follow-up | 2
Not completed — Investigator Decision | 1

BASELINE CHARACTERISTICS:
Population: SP included all participants who were enrolled and received at least one dose of study product.
Groups:
- Minoxidil 5% Foam and Botanical Hair Solution: Participant received minoxidil 2% solution 1 mL on the scalp in the hair loss area and botanical hair solution (5-10 sprays) for women on entire scalp twice per day for up to 12 weeks.
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 5
  Race: Black or African American | 12
  Race: Hispanic or Latino | 11
  Race: White | 31
  Race: Multi-Racial | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. I - Always bums; never tans II - Bums easily; tans minimally III - Burns moderately; tans gradually to light brown IV - Burns minimally; tans well to moderate brown V - Rarely burns; tans profusely to dark brown VI - Never bums; tans profusely to black.
  Participants
    II | 15
    III | 17
    IV | 21
    V | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Investigator's Rating of Global Photographs at Week 12
Description: The Investigator or a trained grader rated each participant's standardized global photographs for improvement from baseline for parameters like hair thinning, hair growth, impression of scalp hair coverage and overall perception of treatment benefit using a 1-to-7-point Likert scale. The score on the scale ranged from 1 (minimum) to 7 (maximum), that is, (1) Entirely Disagree; (2) Mostly Disagree; (3) Somewhat Disagree; (4) Neither Agree nor Disagree; (5) Somewhat Agree; (6) Mostly Agree; (7) Entirely Agree.
Time Frame: At Week 12
Population: ITT population included all participants who were randomized and have at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 54
Score on a scale
  Hair Thinning | 4.9 (0.9)
  Hair Growth | 4.9 (0.8)
  Impression of scalp hair coverage | 4.8 (0.8)
  Overall perception of treatment benefit | 5.0 (0.9)

2. Secondary Outcome: Change From Baseline in Participant Rating at Week 12
Description: Participants rated the parameters like appearance of hair, growth of hair, satisfaction with Hairline at the front of the head, satisfaction with hair on the top of the head and satisfaction with hair overall as an overall improvement from the baseline by conducting their own assessments by looking in a mirror and evaluating improvement from baseline using a 1 to 7-point Likert scale. The scores on the scale ranged from 1 (minimum) to 7 (maximum), that is, (1) Entirely Disagree; (2) Mostly Disagree; (3) Somewhat Disagree; (4) Neither Agree nor Disagree; (5) Somewhat Agree; (6) Mostly Agree; (7) Entirely Agree.
Time Frame: At Week 12
Population: ITT population included all participants who were randomized and had at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 54
Score on a scale
  Appearance of hair | 5.6 (1.3)
  Growth of hair | 5.4 (1.5)
  Satisfaction with hairline at the front of the head | 5.1 (1.5)
  Satisfaction with hair on the top of the head | 5.1 (1.5)
  Satisfaction with hair overall as an overall improvement from the baseline | 5.5 (1.5)

3. Secondary Outcome: Mean Change From Baseline in Shed Hair Count
Description: Participants collected their hair full day, including after combing and hair-washing. Participants turned in these hair collections at each visit. The results were averaged weekly. Mean change from baseline in hair wash/shed hair count was reported at week 12.
Time Frame: At Week 12
Population: The ITT population included all participants who were randomized and had at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Shed Hair Count
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 54
Shed Hair Count | 4.9 (121.8)

4. Secondary Outcome: Number of Participants in Each Response Category Based on Subject Satisfaction Questionnaire
Description: Participant satisfaction with the treatment experience data was collected via a written questionnaire This questionnaire composed of 5-point Likert scale questions, as well as free-text responses. Participants were asked to determine overall satisfaction with the treatment. The choices were: 1-2 = Agree; 4-5 = Disagree; 3 = Neutral.
Time Frame: At Week 4, 6 and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 54
Participants
  I have noticed an improvement in the appearance of my hair (At Week 4): Agree | 27
  I have noticed an improvement in the appearance of my hair (At Week 4): Disagree | 13
  I have noticed an improvement in the appearance of my hair (At Week 4): Neutral | 14
  I have noticed an improvement in the appearance of my hair (At Week 6): Agree | 37
  I have noticed an improvement in the appearance of my hair (At Week 6): Disagree | 9
  I have noticed an improvement in the appearance of my hair (At Week 6): Neutral | 8
  I have noticed an improvement in the appearance of my hair (At Week 12): Agree | 45
  I have noticed an improvement in the appearance of my hair (At Week 12): Disagree | 4
  I have noticed an improvement in the appearance of my hair (At Week 12): Neutral | 5
  This Regimen provides thicker looking hair (At Week 4): Agree | 25
  This Regimen provides thicker looking hair (At Week 4): Disagree | 15
  This Regimen provides thicker looking hair (At Week 4): Neutral | 14
  This Regimen provides thicker looking hair (At Week 6): Agree | 38
  This Regimen provides thicker looking hair (At Week 6): Disagree | 10
  This Regimen provides thicker looking hair (At Week 6): Neutral | 6
  My hair looks fuller (At Week 4): Agree | 25
  My hair looks fuller (At Week 4): Disagree | 16
  My hair looks fuller (At Week 4): Neutral | 13
  My hair looks fuller (At Week 6): Agree | 35
  My hair looks fuller (At Week 6): Disagree | 9
  My hair looks fuller (At Week 6): Neutral | 10
  My hair looks noticeably fuller (At Week 12): number analyzed (Participants) | 52
  My hair looks noticeably fuller (At Week 12): Agree | 38
  My hair looks noticeably fuller (At Week 12): Disagree | 8
  My hair looks noticeably fuller (At Week 12): Neutral | 6
  This Regimen provides healthier looking hair (At Week 4): Agree | 26
  This Regimen provides healthier looking hair (At Week 4): Disagree | 12
  This Regimen provides healthier looking hair (At Week 4): Neutral | 16
  This Regimen provides healthier looking hair (At Week 6): Agree | 31
  This Regimen provides healthier looking hair (At Week 6): Disagree | 8
  This Regimen provides healthier looking hair (At Week 6): Neutral | 15
  I am happy with the appearance of hair (At Week 4): Agree | 24
  I am happy with the appearance of hair (At Week 4): Disagree | 17
  I am happy with the appearance of hair (At Week 4): Neutral | 13
  I am happy with the appearance of hair (At Week 6): Agree | 31
  I am happy with the appearance of hair (At Week 6): Disagree | 12
  I am happy with the appearance of hair (At Week 6): Neutral | 11
  This Regimen improves my hair volume (At Week 4): Agree | 24
  This Regimen improves my hair volume (At Week 4): Disagree | 18
  This Regimen improves my hair volume (At Week 4): Neutral | 12
  This Regimen improves my hair volume (At Week 6): Agree | 35
  This Regimen improves my hair volume (At Week 6): Disagree | 8
  This Regimen improves my hair volume (At Week 6): Neutral | 11
  This Regimen improves my hair volume (At Week 12): Agree | 43
  This Regimen improves my hair volume (At Week 12): Disagree | 5
  This Regimen improves my hair volume (At Week 12): Neutral | 6
  This Regimen improves my hair texture (At Week 4): Agree | 22
  This Regimen improves my hair texture (At Week 4): Disagree | 17
  This Regimen improves my hair texture (At Week 4): Neutral | 15
  This Regimen improves my hair texture (At Week 6): Agree | 28
  This Regimen improves my hair texture (At Week 6): Disagree | 10
  This Regimen improves my hair texture (At Week 6): Neutral | 16
  This Regimen improves my hair texture (At Week 12): Agree | 36
  This Regimen improves my hair texture (At Week 12): Disagree | 10
  This Regimen improves my hair texture (At Week 12): Neutral | 8
  I have noticed an improvement in my hair quality (At Week 4): Agree | 26
  I have noticed an improvement in my hair quality (At Week 4): Disagree | 12
  I have noticed an improvement in my hair quality (At Week 4): Neutral | 16
  I have noticed an improvement in my hair quality (At Week 6): Agree | 35
  I have noticed an improvement in my hair quality (At Week 6): Disagree | 6
  I have noticed an improvement in my hair quality (At Week 6): Neutral | 13
  I have noticed an improvement in my hair quality (At Week 12): Agree | 41
  I have noticed an improvement in my hair quality (At Week 12): Disagree | 7
  I have noticed an improvement in my hair quality (At Week 12): Neutral | 6
  My scalp feels better since beginning this Regimen (At Week 4): Agree | 24
  My scalp feels better since beginning this Regimen (At Week 4): Disagree | 13
  My scalp feels better since beginning this Regimen (At Week 4): Neutral | 17
  My scalp feels better since beginning this Regimen (At Week 6): Agree | 27
  My scalp feels better since beginning this Regimen (At Week 6): Disagree | 6
  My scalp feels better since beginning this Regimen (At Week 6): Neutral | 21
  My hair looks stronger (At Week 4): Agree | 29
  My hair looks stronger (At Week 4): Disagree | 10
  My hair looks stronger (At Week 4): Neutral | 15
  My hair looks stronger (At Week 6): Agree | 35
  My hair looks stronger (At Week 6): Disagree | 8
  My hair looks stronger (At Week 6): Neutral | 11
  My hair looks stronger (At Week 12): Agree | 43
  My hair looks stronger (At Week 12): Disagree | 6
  My hair looks stronger (At Week 12): Neutral | 5
  I like the Regimen I used in this study (At Week 12): number analyzed (Participants) | 52
  I like the Regimen I used in this study (At Week 12): Agree | 43
  I like the Regimen I used in this study (At Week 12): Disagree | 5
  I like the Regimen I used in this study (At Week 12): Neutral | 4
  I received compliments from friends and family members about my hair (At Week 12): number analyzed (Participants) | 52
  I received compliments from friends and family members about my hair (At Week 12): Agree | 23
  I received compliments from friends and family members about my hair (At Week 12): Disagree | 16
  I received compliments from friends and family members about my hair (At Week 12): Neutral | 13
  I would recommend this Regimen to others (At Week 12): number analyzed (Participants) | 52
  I would recommend this Regimen to others (At Week 12): Agree | 42
  I would recommend this Regimen to others (At Week 12): Disagree | 6
  I would recommend this Regimen to others (At Week 12): Neutral | 4
  I feel younger (At Week 12): number analyzed (Participants) | 52
  I feel younger (At Week 12): Agree | 23
  I feel younger (At Week 12): Disagree | 10
  I feel younger (At Week 12): Neutral | 19
  I thought this Regimen did better than my previous hair thinning products (At Week 12): number analyzed (Participants) | 52
  I thought this Regimen did better than my previous hair thinning products (At Week 12): Agree | 23
  I thought this Regimen did better than my previous hair thinning products (At Week 12): Disagree | 8
  I thought this Regimen did better than my previous hair thinning products (At Week 12): Neutral | 21
  I feel more attractive (At Week 12): number analyzed (Participants) | 52
  I feel more attractive (At Week 12): Agree | 33
  I feel more attractive (At Week 12): Disagree | 11
  I feel more attractive (At Week 12): Neutral | 8
  I feel more sociable (At Week 12): number analyzed (Participants) | 52
  I feel more sociable (At Week 12): Agree | 26
  I feel more sociable (At Week 12): Disagree | 11
  I feel more sociable (At Week 12): Neutral | 15
  I feel more confident (At Week 12): number analyzed (Participants) | 52
  I feel more confident (At Week 12): Agree | 31
  I feel more confident (At Week 12): Disagree | 9
  I feel more confident (At Week 12): Neutral | 12
  I would purchase this Regimen (At Week 12): number analyzed (Participants) | 52
  I would purchase this Regimen (At Week 12): Agree | 40
  I would purchase this Regimen (At Week 12): Disagree | 6
  I would purchase this Regimen (At Week 12): Neutral | 6
  My hair looks heathier (At Week 12): number analyzed (Participants) | 52
  My hair looks heathier (At Week 12): Agree | 43
  My hair looks heathier (At Week 12): Disagree | 5
  My hair looks heathier (At Week 12): Neutral | 4

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs were defined as any untoward medical occurrence associated with the use of a study product in humans, whether or not considered study product related. An AE could be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study product and would not imply any judgment about causality. An AE could arise with any use of the study product and with any route of administration, formulation, or dose, including an overdose. Thus any new sign, symptom or disease, or clinically significant increase in the intensity of an existing sign, or symptom would be considered as an AE. Any new clinically relevant sign or symptom suffered by the participant, which appeared after the study procedures was reported as an AE. Any worsening in scalp dryness or itch score from baseline was also reported as an AE. The Investigator or designee had the final authorization to determine if a reaction was considered an AE.
Time Frame: From start of study drug administration up to Week 12
Population: SP included all participants who were enrolled and received at least one dose of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
Number analyzed (Participants) | 60
Participants | 2

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 12
Description: SP included all participants who were enrolled and received at least one dose of study product.
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 4/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minoxidil 5% Foam and Botanical Hair Solution (N=60)
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Influenza (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other